CLINICAL TRIAL: NCT07000539
Title: Prospective Single-center Diagnostic Parallel-group Study to Determine the Minimal Dose of Indocyanine Green to Observe Vascular Perfussion in Revisional Bariatric Surgery.
Brief Title: Indocyanine Green Fluorescence Angiography (ICG-FA) in Revisional Bariatric Surgery
Acronym: BariGreen
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Collaborators: Bariatric Medical Center (Unknown)
Responsible Party: Principal Investigator, : Manuel Alberto Guerrero Gutierrez, Study Director, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: CEI-001-2025042
Record Dates: First submitted 2025-05-24; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Bariatric Surgery
Keywords: bariatric surgery; indocyanine green; vascular; weight loss surgery; Intraoperative Complications; Postoperative Complications
MeSH Terms: conditions — Obesity; Intraoperative Complications; Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Group assignment is centrally managed. Participants are blinded under anesthesia, with no awareness of group assignment. The anesthesiologist knows the dose but is blinded to outcomes and conceals the dose from surgeons. Data collectors and laboratory technicians are not informed of group assignment or study purpose. Adjudicators of outcomes, not involved in surgery, will assess postoperative videos blinded to patient characteristics and knowing only the timing of drug administration. Data analysts and the data safety monitoring committee use coded identifiers to remain blinded to group assignments. The manuscript's results will be written blinded, after which codes will be replaced for actual doses to interpret and discuss the findings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- indocyanine green (5 mg) (Active Comparator): Participants in this arm will receive a single 5 mg intravenous dose of indocyanine green (ICG) during surgery, diluted in 10 mL of sterile saline, followed by a 20 mL saline flush. ICG angiography will be performed using a near-infrared (NIR) fluorescence imaging system (Stryker® 1688 4K laparoscopic camera or da Vinci Xi Firefly®). Imaging will begin immediately before ICG administration and will include a minimal 120 seconds focused on the pouch or duodenal area and the anastomosis. The camera will be positioned at a fixed 5 cm distance and 30° angle. All other surgical procedures will be conducted according to standard of care.
  Interventions: Diagnostic Test: Indocyanine Green Angiogram
- indocyanine green (7.5 mg) (Active Comparator): Participants in this arm will receive a single 7.5 mg intravenous dose of indocyanine green (ICG) during surgery, diluted in 10 mL of sterile saline, followed by a 20 mL saline flush. ICG angiography will be performed using a near-infrared (NIR) fluorescence imaging system (Stryker® 1688 4K laparoscopic camera or da Vinci Xi Firefly®). Imaging will begin immediately before ICG administration and will include a minimal 120 seconds focused on the pouch or duodenal area and the anastomosis. The camera will be positioned at a fixed 5 cm distance and 30° angle. All other surgical procedures will be conducted according to standard of care.
  Interventions: Diagnostic Test: Indocyanine Green Angiogram
- indocyanine green (10 mg) (Active Comparator): Participants in this arm will receive a single 10 mg intravenous dose of indocyanine green (ICG) during surgery, diluted in 10 mL of sterile saline, followed by a 20 mL saline flush. ICG angiography will be performed using a near-infrared (NIR) fluorescence imaging system (Stryker® 1688 4K laparoscopic camera or da Vinci Xi Firefly®). Imaging will begin immediately before ICG administration and will include a minimal 120 seconds focused on the pouch or duodenal area and the anastomosis. The camera will be positioned at a fixed 5 cm distance and 30° angle. All other surgical procedures will be conducted according to standard of care.
  Interventions: Diagnostic Test: Indocyanine Green Angiogram

INTERVENTIONS:
Diagnostic Test: Indocyanine Green Angiogram — Three different doses of indocyanin green will be compared (5 mg, 7.5 mg, and 10 mg). These doses are within the range of currently recommended doses by the International Society for Fluorescence Guided Surgery (ISFGS) for bariatric surgery.
  Other Names: ICG-FA; Indocyanine green fluorescence angiography

SUMMARY:
This study will compare different doses of a green fluorescent product that is administered during weight loss surgery in order to observe where blood vessels are located. There is uncertainty around the optimal dose of this product for patients with obesity, so this study will aim to study if the dose in the minimal range recommended by international guidelines is sufficient for most patients or if higher doses are needed with increasing body mass index.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of obesity with a BMI ≥ 30 kg/m²
* Scheduled for revisional bariatric surgery

Exclusion Criteria:

* Allergy to iodides.
* Anticoagulation with products containing sodium bisulfite (due to the risk of ICG-FA inactivation).
* Use of radioactive iodine studies within the past 7 days.
* Pregnant, breastfeeding, or planning to become pregnant within the next year (due to unknown teratogenic or fertility effects of ICG-FA).
* History of liver disease or laboratory findings suggestive of moderate to severe hepatic disease: total bilirubin >1.5 times the upper limit of normal (ULN), or any elevation of aspartate aminotransferase (AST) above ULN.
* Participants who withdraw their consent to participate in the study (elimination criterion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Time to Fluorescence Detection | Intraoperative (within 5 minutes post-injection)
  Time (in seconds) from intravenous injection of indocyanine green (ICG) to the first visual detection of fluorescence in the surgical field, as captured using near-infrared fluorescence imaging. Assessed at four time points (30s, 60s, 90s, 120s) post-injection. Timing will be standardized from injection to image capture. Time point of first visible fluorescence will be recorded by blinded assessors.

SECONDARY OUTCOMES:
Regional Tissue Perfusion by Anatomical Zone | Intraoperative
  Fluorescence signal intensity and timing will be recorded for predefined anatomical zones based on vascular supply in the gastric pouch and duodenal stump. Zones are classified as Zone 1 (proximal/cardial), Zone 2 (mid/corporal), Zone 3 (distal/anastomotic) for the pouch, and Zone 1 (pyloric transition), Zone 2 (suprapancreatic duodenum), and Zone 3 (distal duodenum) for the duodenum. Signal quality will be scored (e.g., adequate/inadequate) and recorded for each zone.
Change in Surgical Strategy Based on ICG-FA | Intraoperative
  Proportion of cases in which surgical plans were modified intraoperatively (e.g., change in site of anastomosis, reinforcement, or tissue resection) based on ICG perfusion findings.
Adverse Events Related to ICG Use | Within 48 hours postoperatively
  Number and type of adverse events related to ICG administration, including allergic reactions (e.g., rash, anaphylaxis) or abnormal elevations in liver enzymes (AST, ALT, bilirubin) postoperatively.
Postoperative Complications | 30 days postoperatively
  Incidence of postoperative complications within 30 days, including anastomotic leak, infection, bleeding, reoperation, or readmission.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Medico Bariatrico, Tijuana, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data will be deposited and made available through an open acess data repository (i.e., Harvard Dataverse). Any potentially sensitive patient-identifying data will either not be released or will undergo minimization and aggregation/abstraction procedures to reduce participant identification risk. Informed consent forms will indicate that a minimal risk of re-identification cannot be excluded despite all these participant data protection methods, in compliance with current IPD sharing recommendations.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting information will be made available with the final original research article, which will be made available as a preprint within a maximum 1-year term after the study conclusion date. This report will be subsequently sent for publication in a peer-reviewed journal. Other pre-specified outcomes may be reported in separate publication after the main research article, reason why the indicated time frame does not apply for such outcomes. There i
Access Criteria: No data and supporting information access restrictions are anticipated, as these will be deposited in open access repositories (i.e., Harvard Dataverse, Open Science Framework, Zenodo).